CLINICAL TRIAL: NCT03061110
Title: Evaluation of the Use of the Tissue Genesis® Icellator Cell Isolation System® ("Icellator") Autologous Adipose Stromal Vascular Fraction Cells as a Treatment for Post-Irradiated Induced Xerostomia in Head and Neck Cancer Patients
Brief Title: Stromal Vascular Fraction for Treatment of Xerostomia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Internal funding not awarded.
Sponsor: Midwestern Regional Medical Center (Other)
Responsible Party: Principal Investigator, Stephen Ray, MD, Surgeon, Midwestern Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MZ2017003
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Xerostomia Due to Radiotherapy (Disorder)
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to usual care (palliation of symptoms) or injection of stromal vascular fraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Active Comparator): Subjects in the Usual Care arm will receive typical therapies to manage the symptoms of dry mouth including but not limited to: chewing gum, sucking sugar-free candy, sipping water, mouth rinses and over-the-counter artificial saliva preparations.
  Interventions: Other: Usual Care
- Stromal Vascular Fraction (Experimental): Subjects in the Stromal Vascular Fraction arm will receive single injections into each of the six (6) peri-oral salivary glands (parotid, submandibular, sublingual).
  Interventions: Biological: Stromal Vascular Fraction

INTERVENTIONS:
Biological: Stromal Vascular Fraction — Stromal Vascular Fraction will be produced from the subject's own adipose tissue by the Tissue Genesis Icellator device.
  Other Names: Adipose-Derived Stem Cells
  Arms: Stromal Vascular Fraction
Other: Usual Care — Usual care will include over-the-counter and prescription methods to treat xerostomia.
  Other Names: Standard of Care
  Arms: Usual Care

SUMMARY:
Prospective, single center, double armed, randomized treatment with observation only (standard of care) control group. Subjects receiving study treatment will have 6 months of study follow-up. Stromal vascular fraction (SVF), an adipose-derived tissue preparation, will be injected into salivary glands to determine safety and efficacy to restore saliva production in head and neck cancer patients with chronic xerostomia resulting from radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects are both eligible
* Subjects must be 21 years of age or older
* History of treated Head and Neck Cancer, no evidence of active cancer at the time of the study
* Original tumor not located adjacent to the parotid or sub-mandibular glands
* Diagnosis of radiation-induced xerostomia
* study is fully explained
* Females of child bearing potential agree to use acceptable methods of contraception through 6 month study follow-up.
* No current malignancy or history of previous malignancy within the last five years, other than the head and neck cancer, with the exception of adequately treated non-abdominal, non-melanoma cutaneous carcinoma (basal cell or squamous cell carcinoma of the skin)
* Willing to undergo a minor surgical procedure (small-volume liposuction, totaling approximately 60-120cc) and a single treatment of an injection of approximately 30ml of autologous Stromal Vascular Fraction taking approximately 10 minutes
* Abdominal area amenable to liposuction of at least 60-120cc of adipose tissue based on Investigator(s) examination
* Willing to be available for all baseline, treatment and follow-up examinations required by protocol
* Willing to forego participation in any other study throughout the duration of this study unless receiving prior approval by Investigator

Exclusion Criteria:

* Patients taking immunosuppressive therapy in the prior 3 months
* Autoimmune disorders
* Patients who are pregnant or currently breast-feeding children
* Patients participating in a study of an experimental drug or medical device within 60 days of study entry
* Uncontrolled hypertension
* Reported unstable cardiovascular disease (e.g., unstable angina, myocardial infarction within past 6 months, cardiac failure or life-threatening arrhythmia, congestive heart failure) or symptomatic postural hypotension within 6 months before screening
* Hemoglobin A1c > 8% within 8 weeks prior to study treatment
* Current use of steroids or immunosuppressant therapies
* Any other condition, which, in the opinion of the Investigator, would contraindicate treatment, affect compliance, interfere with study evaluations, limit study participation, or confound the interpretation of study results
* History of Sjogren's Syndrome or related autoimmune disease.
* Taking medication for which xerostomia is a known major side effect

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2020-12-28 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute Safety Profile (Reported Adverse Events graded according to CTCAE guidelines) | 72 hours
  Reported Adverse Events graded according to CTCAE guidelines will be recorded starting at or after the time of injection and at or before 72 hours post injection.

SECONDARY OUTCOMES:
Chronic Safety Profile (Reported Adverse Events graded according to Common Terminology Criteria for Adverse Events (CTCAE) guidelines) | Months 3, 6 and 12 after Day 0 (date of injection)
  Reported Adverse Events graded according to Common Terminology Criteria for Adverse Events (CTCAE) guidelines will be recorded starting on Day 0 (day of SVF injection) and ending at 12 months.
Unstimulated Saliva Production | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Rate of saliva production over a 5-minute period. (g/minute)
Stimulated Saliva Production | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Rate of saliva production while chewing gum over a 5-minute period. (g/minute)
University of Rotterdam Hospital Xerostomia Questionnaire- "How severe is your dry mouth problem?" | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score calculated from patient-reported survey (Likert Scale; 1 = Normal; 2 = somewhat more complaints than before radiation therapy; 3 = considerable more complaints than before radiation therapy; and 4 = Permanent complaints of a very dry mouth)
University of Rotterdam Hospital Xerostomia Questionnaire - "Under which circumstances does the dry mouth problem occur? (In the open air) | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Incidence of each indication calculated from categorical patient-reported survey (Yes, No, Not Applicable)
University of Rotterdam Hospital Xerostomia Questionnaire - "Under which circumstances does the dry mouth problem occur? (In the open air in case of wind and cold) | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Incidence of each indication calculated from categorical patient-reported survey (Yes, No, Not Applicable)
University of Rotterdam Hospital Xerostomia Questionnaire - "Under which circumstances does the dry mouth problem occur? (In air-conditioned spaces) | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Incidence of each indication calculated from categorical patient-reported survey (Yes, No, Not Applicable)
University of Rotterdam Hospital Xerostomia Questionnaire - "Under which circumstances does the dry mouth problem occur? (Especially dry mouth during daytime) | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Incidence of each indication calculated from categorical patient-reported survey (Yes, No, Not Applicable)
University of Rotterdam Hospital Xerostomia Questionnaire - "Under which circumstances does the dry mouth problem occur? (Especially dry mouth at nighttime) | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Incidence of each indication calculated from categorical patient-reported survey (Yes, No, Not Applicable)
University of Rotterdam Hospital Xerostomia Questionnaire - "Under which circumstances does the dry mouth problem occur? (Always dry mouth night and day) | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Incidence of each indication calculated from categorical patient-reported survey (Yes, No, Not Applicable)
University of Rotterdam Hospital Xerostomia Questionnaire - "Under which circumstances does the dry mouth problem occur? (Especially bother of the dry mouth during meals) | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Incidence of each indication calculated from categorical patient-reported survey (Yes, No, Not Applicable)
University of Rotterdam Hospital Xerostomia Questionnaire- "How often do you wake up at night because of a dry mouth?" | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Number of events as reported by patient (Number)
University of Rotterdam Hospital Xerostomia Questionnaire - "How would you describe the quality of your saliva?" | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score calculated from patient-reported survey (Likert Scale; 1 = Normal, watery fluid; 2 = Normal watery but too little volume; 3 = Sticky saliva; and 4 = No saliva at all)
University of Rotterdam Hospital Xerostomia Questionnaire - "Do you have difficulties with speech because of the dry mouth?" | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score calculated from patient-reported survey (Likert Scale; 1 = No problems; unchanged with respect to situation before radiation therapy; 2 = Occasionally some difficulty with speech; 3 = Frequently speech problems; 4 = always difficulties with speech; and 5= always major speech problems)
University of Rotterdam Hospital Xerostomia Questionnaire - "Do you need to sip water to facilitate speech?" | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score calculated from patient-reported survey (Likert Scale; 1 = Never; 2 = Occasionally; 3 = Frequently; 4 = Always; and 5= Even have to interrupt speaking to take a sip of water)
University of Rotterdam Hospital Xerostomia Questionnaire - "Is swallowing changed because of the dry mouth problem?" | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score calculated from patient-reported survey (Likert Scale; 1 = No problems; unchanged with respect to situation before radiation therapy; 2 = Occasionally some difficulty with swallowing; 3 = Frequently problems with swallowing; 4 = Always swallowing difficulties; and 5 = Swallowing is seriously impaired because of the dry mouth problem)
University of Rotterdam Hospital Xerostomia Questionnaire - "Has the dry mouth a negative influence on chewing?" | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score calculated from patient-reported survey (Likert Scale; 1 = No change in chewing capability; 2 = Some difficulty with chewing; 3 = Frequently difficulties with chewing; 4 = Always difficulties with chewing; 5 = Chewing is seriously hampered because of the dry mouth problem)
University of Rotterdam Hospital Xerostomia Questionnaire - "Do you need to sip water to facilitate eating?" | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score calculated from patient-reported survey (Likert Scale; 1 = No never; 2 = Sometimes, depending on the quality of the food; 3 = Frequently; more often than before radiation therapy; and 4 = Always need to take a sip of water/ fluid with every bite of food)
University of Rotterdam Hospital Xerostomia Questionnaire - "Did you change your feeding habits?" | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score calculated from patient-reported survey (Likert Scale; 1 = No change; 2 = Minor changes, such as avoiding some products; 3 = Can eat only mashed food; 4 = Can eat only liquid food; and 5= Tube feeding)
University of Rotterdam Hospital Xerostomia Questionnaire - "Do you have painful, dry, or crusted lips?" | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score calculated from patient-reported survey (Likert Scale; 1 = Never; 2 = Sometimes, depending on the weather and environmental circumstances; 3 = Frequently; and 4 = Always, day and night)
University of Rotterdam Hospital Xerostomia Questionnaire - "Do you need to carry a bottle of fluid with you when leaving home?" | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score calculated from patient-reported survey (Likert Scale; 1 = Never 2 = Occasionally; 3 = Frequently; 4 = Very often; and 5 = Always)
University of Rotterdam Hospital Xerostomia Questionnaire - "Do you have a sore or painful mouth?" | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score calculated from patient-reported survey (Likert Scale; 1 = Never 2 = Occasionally; 3 = Frequently; 4 = Very often; and 5 = Always)
University of Rotterdam Hospital Xerostomia Questionnaire - "Did your taste change?" | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score calculated from patient-reported survey (Likert Scale; 1 = No change; normal taste sensation; 2 = Some reduction in taste discrimination and sensation; 3 = Considerable change in taste; 4 = No taste sensation at all; and 5 = Always a bad taste in the mouth)
University of Rotterdam Hospital Xerostomia Questionnaire - "Do you often have an infected oral mucosa or irritated gums?" | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Incidence of each indication calculated from categorical patient-reported survey (Yes, No, Not Applicable)
University of Rotterdam Hospital Xerostomia Questionnaire - "Did your teeth deteriorate after radiation therapy?" | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score calculated from patient-reported survey (Likert Scale; 1 = never; 2 = Occasionally; 3 = Frequently; and 4 = Very often)
University of Rotterdam Hospital Xerostomia Questionnaire - Overall Xerostomia Index | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Overall Xerostomia Index is calculated from the first three questions of the Questionnaire [I = (Q1 x 15.8) + (Q2 x 8.5) + (Q3 x 5.9) - 33.2; where Qn = score of that question.]
University of Michigan Xerostomia-Related Quality of Life Scale - Physical Functioning | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score calculated from patient-reported survey (Likert Scale; 0=Best Functioning to 4=Worst Functioning)
University of Michigan Xerostomia-Related Quality of Life Scale - Pain/Discomfort | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score calculated from patient-reported survey (Likert Scale; 0=No Pain to 4=Worst Pain)
University of Michigan Xerostomia-Related Quality of Life Scale - Personal/Psychological Functioning | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score calculated from patient-reported survey (Likert Scale; 0=Best Functioning to 4=Worst Functioning)
University of Michigan Xerostomia-Related Quality of Life Scale - Social Functioning | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score between Baseline and 3 months calculated from patient-reported survey (Likert Scale; 0=Best Functioning to 4=Worst Functioning)
Late Effects Normal Tissue-Subjective Objective Management Analytica (LENT-SOMA) survey | Assessed at Baseline and 3 months, 6 months and 12 months after Baseline
  Mean score calculated from patient-reported survey (Likert Scale; 1=Best Functioning to 4=Worst Functioning)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ray, MD, Principal Investigator — Midwestern Regional Medical Center
Locations (1):
- Midwestern Regional Medical Center, Zion, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided